CLINICAL TRIAL: NCT00847704
Title: Clinic-Based Ames Treatment of the Lower Extremity in Chronic Stroke Subjects
Brief Title: Clinic-Based AMES Treatment of Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding not available.
Sponsor: Oregon Health and Science University (Other)
Collaborators: AMES Technology (Industry)
Responsible Party: Principal Investigator, Paul J. Cordo, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 4005; NCT00600184 (obsolete NCT alias)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Stroke; Rehabilitation; Robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test treatment group (Experimental): Device: Assisted movement and enhanced sensation
  Interventions: Device: Assisted movement and enhanced sensation

INTERVENTIONS:
Device: Assisted movement and enhanced sensation — Each subject will be tested before, after the 10 week treatment period and then 3 months later. Treatment sessions will occur 3 times per week and last approximately 30 minutes per treatment. The device will measure 3 of the functional tests prior to each treatment session.

SUMMARY:
This study investigates whether assisted movement with biofeedback and muscle vibration applied to the lower limb reduces impairment and improves gait.

DETAILED DESCRIPTION:
The hypothesis of this study is that chronic stroke survivors, more than one year post-stroke, with a motor problems in the lower extremity will be able to walk and move the affected leg better after 30 treatments with a new robotic therapy device, the AMES device. The device rotates the ankle while vibrators stimulate the tendons attached to muscles that move the ankle. Testing will be done before, during and after the treatments to determine response to the therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months post-stroke
* Cognitively and behaviorally capable of complying with the regimen
* Functioning proprioception
* Less than 50% of normal strength in the affected ankle, but able to stand with or without assistive devices

Exclusion Criteria:

* Fractures of treated limb resulting in loss of range of motion
* Spinal cord injury
* Deep vein thrombosis
* Peripheral nerve injury or neuropathy in the limb affected with motor disability
* Osteoarthritis limiting range of motion
* Skin condition not tolerant of device
* Progressive neurodegenerative disorder
* Uncontrolled seizure disorder
* Botox treatment within the last 5 months
* Baclofen pump

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Cordo, PhD, Principal Investigator — AMES Technology Inc./Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Cordo P, Lutsep H, Cordo L, Wright WG, Cacciatore T, Skoss R. Assisted movement with enhanced sensation (AMES): coupling motor and sensory to remediate motor deficits in chronic stroke patients. Neurorehabil Neural Repair. 2009 Jan;23(1):67-77. doi: 10.1177/1545968308317437. Epub 2008 Jul 21. PMID 18645190

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: Device: Assisted movement and enhanced sensation
Period: Overall Study
Arm/Group | Test Group
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Stroke >1 yr prior to enrollment Able to stand independently <50% normal strength in affected leg Functioning proprioception in affected leg
Groups:
- Test Group: Device: Assisted movement and enhanced sensation
  Assisted movement and enhanced sensation: Each subject will be tested before, after the 10 week treatment period and then 3 months later. Treatment sessions will occur 3 times per week and last approximately 30 minutes per treatment. The device will measure 3 of the functional tests prior to each treatment session.
  Assisted movement and enhanced sensation: Thirty treatment sessions on the AMES device, each session 30 minutes of cyclic rotation of the ankle with tendon vibration. Testing before, during, and after treatments to evaluate response to treatments.
Arm/Group | Test Group
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (2.0)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2
Time since stroke [Mean (Standard Deviation); unit: Months] | 113.5 (85.5)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment of the Lower Extremity
Description: Gold standard for motor impairment in individuals with stroke. A scale measuring tone, range-of-motion and synergies of the lower limb with a range of 0-34, higher scores referring to improved motor ability. The assessment includes 7 subscales, the scores of which are summed to arrive at a total score.
Time Frame: Pre-training, After 30 training sessions (8-10 weeks), 3-Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Group: Group receiving AMES therapy
Arm/Group | Test Group
Number analyzed (Participants) | 2
units on a scale
  Baseline | 21.0 (1.0)
  Post-treatment | 19.5 (0.5)
  3 Month Follow-up | 21 (1.0)

2. Secondary Outcome: Timed 10-Meter Walk
Description: Gait Assessment - Time
Time Frame: Pre-training, After 30 training sessions (8-10 weeks), 3-Month Follow-up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Test Group
Number analyzed (Participants) | 2
seconds
  Baseline | 12.465 (0.055)
  Post-treatment | 13.66 (0.34)
  3 Month Follow-up | 13.27 (0.11)

3. Secondary Outcome: Stroke Impact Scale
Description: The Stroke Impact Scale is a self-assessment questionnaire concerning activities of daily living. There are 8 sub-scales, each of which is summed as a raw score (range of 0-100) and then transformed as follows:
  Transformed Scale=[(Actual raw score-lowest possible raw score)/Possible raw score range]x100.
  Thus, the maximum possible score for the entire measure is 800. A higher score indicates a higher level of functioning.
Time Frame: Pre-training, After 30 training sessions (8-10 weeks), 3-Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Group
Number analyzed (Participants) | 2
units on a scale
  Baseline | 234.5 (9.5)
  Post-treatment | 258 (4.0)
  3 Month Follow-up | 251.5 (1.5)

4. Secondary Outcome: Spasticity (Modified Ashworth) Scale
Description: Measure of the total Ashworth scoring for increased muscle tone in the ankle flexors, ankle extensors, knee flexors, and knee extensors in the affected leg of stroke subjects. The scale range is from 0-5, with higher levels representing more exaggerated tone.
Time Frame: Pre-training, After 30 training sessions (8-10 weeks), 3-Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Group
Number analyzed (Participants) | 2
units on a scale
  Baseline | 2.0 (2.0)
  Post-treatment | 0.5 (0.5)
  3 Month Follow-up | 2.0 (1.0)

5. Secondary Outcome: Strength Test
Description: Measurement of ankle dorsiflexion/plantarflexion isometric strength (change-score from average of first 3 training sessions and last 3 training sessions).
Time Frame: First 3 training sessions (week 1-2); Last 3 training sessions (week 9-10)
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Test Group
Number analyzed (Participants) | 2
Newton meters
  Dorsiflexion | 33.7 (41.4)
  Plantarflexion | 31.5 (8.8)

6. Secondary Outcome: Active Motion Test
Description: Tracking task. Active joint position control between dorsiflexion/plantarflexion (change-score from average of first 3 training sessions and last 3 training sessions). The score is based on the amount of time that the participant is able to position the joint in a 3 deg-wide target zone presented on a video screen.
Time Frame: First 3 training sessions (week 1-2); Last 3 training sessions (week 9-10)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Test Group
Number analyzed (Participants) | 2
Seconds | 5.8 (0.2)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Description: Verbal inquiry at the beginning of each training session.
Groups:
- Test Treatment Group: Device: Subjects receiving AMES treatments.
Arm/Group | Test Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Treatment Group (N=3)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Loss of balance during moving

LIMITATIONS AND CAVEATS:
Early termination due to lack of funding lead to only 2 subjects treated and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes